CLINICAL TRIAL: NCT03391544
Title: Rotational Stability of V4C Toric Implantable Contact Lenses After On Axis Implantation Measured With OPD Scan 3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2017-0243
Record Dates: First submitted 2017-12-21; First posted 2018-01-05 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2017-12

CONDITIONS: Myopic Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- V4c toric ICL implantation Group (Experimental): V4c toric ICL implantation Group
  Interventions: Procedure: V4c toric ICL implantation surgery

INTERVENTIONS:
Procedure: V4c toric ICL implantation surgery — The size and power of the V4c toric ICL were determined following the manufacturer's guidelines using a modified vertex formula. Emmetropia was the target refraction following surgery in all cases. Before surgery, three centration points were marked using the slit lamp while the patient, in sitting position, fixated on the center of the slit-lamp beam, which was narrowed as much as possible.

SUMMARY:
The recently introduced toric V4c toric ICL (STAAR Surgical Company, Monrovia, CA, USA) has been designed with a 360-µm central hole to allow aqueous humor to flow without the need for an iridotomy. As far as the investigators certain, there have been not well-established prospective studies on the role of the V4c toric ICL for myopic astigmatism correction. Therefore, the present study aimed to investigate the clinical outcomes and rotational stability and to analyze factors that influence the rotational stability in V4c toric ICL implanted eyes prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-45 years
* Presence of myopia with a manifest refraction spherical equivalent between -5.00 and -20.00 diopters (D)
* Astigmatism between -0.75 and -5.00 D

Exclusion Criteria:

* Previous ocular or intraocular surgery (other than ICL implant)
* Anterior chamber depth from the endothelium < 2.8 mm
* Corneal endothelial cell density < 2000 cells/mm2
* Evidence of acute or chronic corneal infection, corneal inflammation
* Glaucoma, amblyopia, retinal detachment, diabetic retinopathy, macular degeneration, or neuro-ophthalmic disease

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2017-04-28 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Visual outcome | 6 months after the surgery
  Evaluation of logarithm of the minimum angle of resolution (logMAR) uncorrected distance visual acuity (UDVA) and CDVA, manifest refraction, autorefractor-keratometer (ARK-530A; Nidek Co., Ltd.). The change of astigmatism was analyzed by the Alpins method.
Refractive outcome | 6 months after the surgery
  Evaluation of logarithm of the minimum angle of resolution (logMAR) uncorrected distance visual acuity (UDVA) and CDVA, manifest refraction, autorefractor-keratometer (ARK-530A; Nidek Co., Ltd.). The change of astigmatism was analyzed by the Alpins method.

SECONDARY OUTCOMES:
Rotational stability | immediately after the surgery
  Rotational stability of the toric ICL was measured using the OPD-Scan III (NIDEK Co. Ltd., Gamagori, Japan). The rotation was defined as the difference between the intended axis and the achieved axis at each follow-up. Assuming that the adjusted axis was identical to the intended angle, postoperative rotation was automatically measured by determining the angle between the adjusted axis and alignment axis. Each measurement was performed three times by one physician, and the average of the three measurements was used in the analysis.
Rotational stability | 3 months after the surgery
  Rotational stability of the toric ICL was measured using the OPD-Scan III (NIDEK Co. Ltd., Gamagori, Japan). The rotation was defined as the difference between the intended axis and the achieved axis at each follow-up. Assuming that the adjusted axis was identical to the intended angle, postoperative rotation was automatically measured by determining the angle between the adjusted axis and alignment axis. Each measurement was performed three times by one physician, and the average of the three measurements was used in the analysis.
Rotational stability | 6 months after the surgery
  Rotational stability of the toric ICL was measured using the OPD-Scan III (NIDEK Co. Ltd., Gamagori, Japan). The rotation was defined as the difference between the intended axis and the achieved axis at each follow-up. Assuming that the adjusted axis was identical to the intended angle, postoperative rotation was automatically measured by determining the angle between the adjusted axis and alignment axis. Each measurement was performed three times by one physician, and the average of the three measurements was used in the analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No